CLINICAL TRIAL: NCT06606002
Title: The Effectiveness of Group Schema Therapy Utilizing Video Material in the Treatment of Borderline Symptoms in Adolescents: A Randomized and Controlled Intervention Study
Brief Title: The Effectiveness of Group Schema Therapy in the Treatment of Borderline Symptoms in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Principal Investigator, Max Karukivi, Associate Professor, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1709/2024
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Borderline Symptoms; Borderline Personality Disorder
Keywords: adolescents; borderline disorder; schema therapy; randomized controlled study
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group schema therapy (Experimental): The group schema therapy intervention includes 30 group sessions and 8 individual sessions for the participants, and 9 group sessions for the participants' parents.
  Interventions: Behavioral: Group schema therapy
- Control (Active Comparator): Treatment as usual
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: Group schema therapy — Group schema therapy based on the model by Farrell and Shaw, which is complemented with separate group sessions for the participants' parents
  Arms: Group schema therapy
Behavioral: Treatment as Usual (TAU) — TAU typically comprises visits at the outpatient clinic with variable frequency and content
  Arms: Control

SUMMARY:
The goal of this randomized and controlled trial is to assess the effectiveness of group schema therapy in the treatment of adolescents with borderline symptoms. The intervention utilizes self-recorded video material as an experiential method. The intervention comprises 30 group sessions and 8 individual sessions. Additionally, there are group sessions for the participants' parents. Participants in the control group receive treatment as usual.

DETAILED DESCRIPTION:
The goal of this randomized and controlled intervention study is to assess the effectiveness of group schema therapy in the treatment of adolescents with borderline symptoms. Borderline personality disorder (BPD) is a severe and chronic mental health disorder, which features are typically detectable already in adolescence. BPD causes considerable suffering and functional impairment. Treatment recommendations emphasize treating BPD with targeted interventions already in adolescence, but evidence-based treatments in this age group are so far scarce.

The research sample consists of 32 adolescents who participate in a group schema therapy intervention and their 32 controls. The participants are adolescents aged 15-18 who are being treated at the Adolescent Psychiatry Clinic at the Turku University Hospital. The subjects meet at least three diagnostic criteria for BPD based on SCID-II assessment. Adolescents who are at serious suicide risk or with, for example, psychotic symptoms, or another disorder or symptom that endangers commitment to the intervention protocol, are excluded from the study.

The studied intervention is based on Farrell and Shaw's group schema therapy model. The experiential part of the model is strengthened utilizing videos, which are recorded by the participants (VideoTalk). The videos are used to support both individual and group work. The intervention is tailored to be developmentally sensitive for this age group and reinforced with a module to which the participants' parents participate.

The intervention comprises 30 weekly group sessions and 8 individual sessions. Eight adolescents participate in one group, and four groups are carried out during the study. The participants' parents have 9 group sessions, some of which the adolescents also participate in. The duration of the intervention is approximately one year. The control group receives treatment as usual.

Both the intervention and control groups response to the research questionnaires at five time points (baseline, 3 months, 6 months, 12 months, 2 years). The primary response variable is the change in the BPD symptoms between entering the study and the end of the intervention. As secondary response variables, changes in, for example, the participants' early maladaptive schemas, schema modes, and depressive and anxiety symptoms are assessed. After the end of the intervention, the study includes a one-year follow-up period and two years after the intervention, follow-up data is collected from the participants' medical reports. The study also includes qualitative sub-studies.

The intervention groups will be carried out during the years 2025-2027. A new group is always started overlapping with the previous group. Results regarding the primary response variable will be completed at the end of 2027. The entire research material will be completed at the end of 2029.

ELIGIBILITY:
Inclusion Criteria:

* The participant fulfills at least three diagnostic criteria for borderline personality disorder as assessed by means of the SCID-II structured clinical interview
* The participant and the participant's parent(s) are able to commit to the research protocol for the entire duration of the study
* The participant is able to participate in a research intervention in Finnish and fill out the study questionnaires in Finnish

Exclusion Criteria:

* The participant currently has psychotic symptoms or a serious risk of suicide
* The participant has been diagnosed with an intellectual disability or an autism spectrum disorder
* The main clinical diagnosis of the participant is a substance abuse disorder or substance use would endanger commitment to the research intervention
* The participant has another illness or symptom that endangers the participant's ability to complete the study
* The participant receives some other treatment specifically aimed at borderline personality disorder symptoms

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Borderline Symptom List - Short version | From enrollment to the end of treatment at 12 months

SECONDARY OUTCOMES:
Young Schema Questionnaire Short Form 2 -Extended | From enrollment to the end of treatment at 12 months
Schema Mode Inventory | From enrollment to the end of treatment at 12 months
Patient Health Questionnaire-9 | From enrollment to the end of treatment at 12 months
Child and Adolescent Trauma Screen | From enrollment to the end of treatment at 12 months
General Anxiety Disorder-7 | From enrollment to the end of treatment at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Max Karukivi, MD, PhD, Principal Investigator — University of Turku
Locations (1):
- Turku University Hospital, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: No